CLINICAL TRIAL: NCT05885139
Title: The Effects of EXOPULSE Mollii Suit on Motor Functions in Children With Cerebral Palsy (EXOCEP 2 GER)
Brief Title: Exopulse Mollii Suit, Motor Functions & CP Children With Cerebral Palsy
Acronym: EXOCEP2GER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Exoneural Network AB (Industry)
Collaborators: Ottobock SE & Co. KGaA (Unknown); Hannover Medical School (Other); Pohlig GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PS00011278C-001
Record Dates: First submitted 2023-04-20; First posted 2023-06-01 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy; Spasticity; Muscle; Pain Syndrome; Hemiplegia; Diplegia; Tetraplegia; Balance
Keywords: Exopulse; Mollii Suit; Spasticity; Neurostimulation
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Somatoform Disorders; Hemiplegia; Quadriplegia

STUDY DESIGN:
Intervention Model Description: Active Comparator: Active Active sessions will last 1 hour each. The following parameters will be used for electric stimulation: low frequency (20 Hz), low current intensity (2 mA), with a small pulse width of 25-170 microseconds. Sham Comparator: Sham In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Stimulation (Active Comparator): Active sessions will last 1 hour of stimulation per day for 2 weeks. The following parameters will be used for electric stimulation: low frequency (20 Hz), low current intensity (2 mA), with a small pulse width of 25-170 microseconds.
  Interventions: Device: Exopulse Mollii Suit
- Sham Stimulation (Sham Comparator): In the sham condition, subjects will be asked to wear the device for 1 hour per day for 2 weeks. During 1 hour use per day, the actual stimulation will last only 1 minute and then will shut off.
  Interventions: Device: Sham Exopulse Mollii Suit

INTERVENTIONS:
Device: Exopulse Mollii Suit — Exopulse Mollii suits consists of a body Garments (Jacket and Pants) and a control unit. The body Garments (Jacket and Pants) is a suit with 58 embedded electrodes that can stimulate 40 groups of muscles, conductive wires and connectors to a detachable control unit, whose intended purpose is to transmit electric pulses from the control unit to key nerves and corresponding muscle groups throughout the body. The control unit is a battery powered electrical device which sends low intensity electric pulses through connectors to the Body Garments which in turn transmits the pulses from the connectors to key nerves and corresponding muscle groups throughout the body.
  Arms: Active Stimulation
Device: Sham Exopulse Mollii Suit — In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off.
  Arms: Sham Stimulation

SUMMARY:
Cerebral Palsy (CP) is is estimated to be around 1.5-3 per live birth, with prenatal factors accounting for 75% of cases. CP appears in early childhood and persists with age and is characterized by permanent lesions or abnormalities affecting the immature brain. It mainly occurs as a motor system disorder (e.g., abnormal movements or posture) with the presence of hemiplegia, diplegia or tetraplegia, and spastic, dyskinetic or atactic syndromes. .This study will explore the potential clinical benefits of the Molliimethod in children with cerebral palsy. Spasticity impacts balance and mobility, halts the patients quality of life and their ability to perform their activity of daily living, and could also increase the risk of fractures and falls. Available interventions that aim on improving spasticity are facing limitations such as varios side effects. Therefore, developing novel therapies such as the EXOPULSE Mollii Suit could help to overcome such limitations and noninvasively improve balance, mobility, quality of life and reduce spasticity and pain in children with CP.

DETAILED DESCRIPTION:
Cerebral Palsy is a heterogenous group of disorders that was first introduced in the literature in 1843 by Little who described musculoskeletal deformities and spastic limbs in the context of neonatal hypoxia. The clinical classification of CP could be based on several system. For instance, the classification by Balf and Ingram takes into account the type, lesion location and severity of the clinical symptoms, and entails the following CP types that could be further considered as mild, moderate or severe: diplegia, hemiplegia or tetraplegia with the presence of spastic syndromes, dyskinetic syndromes and ataxia. In the context of CP, spasticity is a frequent and debilitating symptom that could occur in 70-89% of individuals. Spasticity could subsequently alter the development of motricity, quality of life, patients' self-es-teem and seems to be associated with several health consequences, namely pain, infections, joint deformities, thrombosis and bedsores. Managing spasticity in CP include the combination of pharmacotherapy, motor rehabilitation, and surgical interventions. It is now widely accepted that spasticity impacts balance and mobility, halts the patients quality of life (e.g., urinary symptoms, sexual dysfunction, mood symptoms, low self-esteem) and their ability to perform their activity of daily living, and could also increase the risk of fractures and falls. The available interventions targeting spasticity are faced with some limitations. For instance, botulinum toxin injection does not seem to improve motor functions and quality of life as well as available oral agents are challenged by their potential side effects. Therefore, developing novel therapies would help to overcome the actual limitations. Transcutaneous Electrical Nerve Stimulation (TENS) has proven some efficacy in spasticity management. However, one should note that practical difficulties could arise when using TENS at home or in clinical practice (i.e., correctly attaching electrodes). To overcome these limitations, the Exopulse Mollii Suit has been developed by Exoneural Network AB (initially Inerventions AB), a Swedish medtech company. It represents an innovative approach for non-invasive electrostimulation to reduce spasticity and improve motor function. Based on the theoretical and practical background outlined above, this study will explore the potential clinical benefits of the Mollii-method in children with cerebral palsy. The overall aim of this study is to evaluate the short-term impact of Exopulse Mollii Suit on balance in pediatric patients with cerebral palsy who are suffering from spasticity as well as assessing the effects of Exopulse Mollii Suit on spasticity, mobility, pain, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they

* are between 5 and 12 years of age.
* have a clinical diagnosis of unilateraal or bilateral spastic CP by birth [15].
* have a PBS score between a minimum of 15 and a maxmimum of 44 points.
* are able to walk freely, with slight limitation or using ancillary equipment's (GMFCS score ≤3) [49].
* are German speakers, able to understand verbal instructions.
* have spasticity with a score of at least 1+ on the MAS

Exclusion Criteria:

Patients will not be included if they

* are included in another research protocol during the study period.
* are unable to undergo clinical procedures for the study purposes due to geographical or social reasons.
* have a cardiac stimulator, a ventriculoperitoneal shunt, intrathecal baclofen pump.
* have a change in their pharmacological therapy over the last three months or are planning to do so during the study.
* suffer from other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain).
* have a body mass index above 35 kg/m2,
* have contraindications to wearing Exopulse Mollii Suit, receive a medical device other than Exopulse Mollii during the study period.
* have received botulinum toxin (botox) therapy in the last 3 months before the start of the study

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Pediatric Balance Scale (PBS) | Visit 1 = Immediately before and after 1h stimulation; Visit 2 = 2 weeks after visit 1; Visit 3 = Immediately before and after 1h stimulation, 4 weeks after visit 1; Visit 4 = 6 weeks after visit 1
  Pediatric patients with CP, the PBS has a minimum detectable change (MDC) of 1.59 for the total score and 0.79 (static) and 0.96 (dynamic) for the subscores. Furthermore, the PBS has a minimally clinically important difference (MCID) for the cohort mentioned of 5.83 for the otal score and 2.92 (static) and 2.92 (dynamic) for the subscores.

SECONDARY OUTCOMES:
Changes in Modified Ashworth Scale (MAS) | Visit 1 = Immediately before and after 1h stimulation; Visit 2 = 2 weeks after visit 1; Visit 3 = Immediately before and after 1h stimulation, 4 weeks after visit 1; Visit 4 = 6 weeks after visit 1
  The modified Ashworth Scale measures spasticity in patients with lesions of the Central Nervous System. It tests resistance to passive movement in a joint with varying degrees of velocity. Scores range from 0-4 with 5 choices. A score of 1 indicates no resistance, and a 5 indicates rigidity.
Changes in Timed Up and Go (TUG) | Visit 1 = Immediately before and after 1h stimulation; Visit 2 = 2 weeks after visit 1; Visit 3 = Immediately before and after 1h stimulation, 4 weeks after visit 1; Visit 4 = 6 weeks after visit 1
  In the chair with his/her back against the chair back. On the command "go", the patient rises from the chair, walks 3Visit 1 = Immediately before and after first 1h stimulation; Visit 2 = 2 weeks after visit 1; Visit 3 = 4 weeks after visit 1. Immediately before and after first 1h stimulation; Visit 4 = 6 weeks after visit 1 meters at a comfortable and safe pace, turns, walks back to the chair and sits down. Timing begins at the instruction "go" and stops when the patient is seated.

OTHER OUTCOMES:
Patient Diary | Visit 1; Visit 2 = 2 weeks after visit 1; Visit 3 = 4 weeks after visit 1. Visit 4 = 6 weeks after visit 1
  4. Patient Diary A patient diary is provided to patiets to record information during the 14-day homeuse phase. If the child is not able to do this him/herself, the parent or cargicer can support this process. The use of the Exopulse Mollii Suit should be recorded, whether the stimulation duration of 1 hour is adhered every day. In addition, comfort/satisfaction, pain/discomfort and possible incidents such as mild adverse events should be documented.
Blinding Questionnaire | Visit 2 = 2 weeks after visit 1; Visit 4 = 6 weeks after visit 1
  Evaluation of patient's blinding to the type of stimulation will be performed by asking for their perception which treatment they received: "(a) Treatment/ (b) Placebo/ (c) I don' know" and "if (c) I don't know" which they would by chance choose "(a) Treatment/ (b) Placebo.
Changes in Functional Gait Assessment (FGA) | Visit 1 = Immediately before and after 1h stimulation; Visit 2 = 2 weeks after visit 1; Visit 3 = Immediately before and after 1h stimulation, 4 weeks after visit 1. ; Visit 4 = 6 weeks after visit 1
  (optional)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Pohlig GmbH, Traunstein, Bavaria
  - Medizinische Hochschule Hannover (MHH), Hanover

IPD SHARING:
Plan to Share IPD: No